CLINICAL TRIAL: NCT01291706
Title: Prospective, Multicentre, Observational Study
Brief Title: Transcranial Doppler on Admission of Patients With Mild to Moderate Traumatic Brain Injury
Acronym: TCD
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: CIC Clinical Investigation Centre Grenoble (Unknown)
Responsible Party: Sponsor
Other Study IDs: DCIC 10 17
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Traumatic Brain Injury
Keywords: Transcranial Doppler; Mild and moderate Traumatic Brain Injury; Neurological deterioration; Brain CT scan
MeSH Terms: conditions — Brain Injuries, Traumatic; Lymphoma, Follicular | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mild TBI with mild lesions on CT scan: Negative predictive value of transcranial doppler for patients with mild to moderate traumatic brain injury and mild brain lesions on initial CT scan (TCDB II)
  Interventions: Device: Transcranial Doppler

INTERVENTIONS:
Device: Transcranial Doppler — Negative predictive value of transcranial doppler in patients with mild to moderate traumatic brain injury

SUMMARY:
Patients with mild to moderate traumatic brain injury (TBI) are at risk for secondary neurological deterioration. Their outcome within the first week after injury could be predicted by clinical signs, brain CT scan and transcranial doppler (TCD) on admission to the emergency room. The investigators aim to evaluate the diagnostic performance of TCD to screen patients presented with mild to moderate TBI and mild lesions on CT scan, i.e., Trauma Coma Data Bank, TCDB classification II. The principal outcome measure is the negative predictive value of TCD.

ELIGIBILITY:
Criteria for inclusion:

* 15 years of age or more
* primary admission for mild TBI (GCS 14-15) or moderate (GCS 9-13) TBI.
* with or without multiple injury.
* with no hemodynamic or respiratory distress: SAP >90mmHg, SPO2 >92%,hemoglobin > 8 g/dl.
* with mild brain lesions on CTscan according to the traumatic coma data bank classification (TCDB) II: diffuse injury with cisterns present and no midline shift, mixed density lesions <25 ml.
* Transcranial Doppler within 8 hours after the trauma.
* patient affiliated to the social security system or equivalent

Criteria for exclusion:

* Severe TBI (GCS<9)
* Penetrating TBI
* patient with no brain CT scan
* patient with normal brain CT scan (TCDB I), or severe brain CT scan (TCDB III-IV)
* Hemodynamic or respiratory distress
* Patient treated with anticoagulants: oral anticoagulant, heparin, anti-platelet agent (except Aspirin)
* previous intracranial surgery
* Patient with sedation and mechanical ventilation
* transcranial Doppler unable
* patient deprived of freedom by judicial or administrative decision
* Follow up at 7 days impossible
* Refusal consent to use data for statistics

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary admission of patients following mild to moderate traumatic brain injury who need exploration with brain CT scan.
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2011-02; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Negative predictive value of transcranial doppler | within the first week after the injury
  Patient with mild to moderate traumatic brain injury (Glasgow Coma Scale 9-15) and a CT scan (TCDB II).TCD is performed within 8 hours after the trauma.
  Aggravation defined by:
  * a decrease in the Glasgow Coma Scale of 2 points or more from the initial value, in the absence of pharmacological sedation.
  * a neurological deterioration sufficient to warrant intervention: mechanical ventilation, sedation, osmotherapy, barbiturates, transfer to more intensive care, or neurosurgical intervention.

SECONDARY OUTCOMES:
the impact of transcranial doppler for initial patient management | within the first week after trauma
  Number of brain CTscan performed within 7 days after the trauma.
  Number of devices inserted to monitor intracranial pressure.
  Secondary admissions to intensive care unit.
  Length of hospital stay.
Secondary neurological aggravation: risk factors and consequences. | neurological outcome on D7 and D28
  Neurological outcome on day 7 and day 28 after trauma, as measured with disability rating scale.
  Number and type of interventions for neurological deterioration

CONTACTS AND LOCATIONS:
Overall Officials: Jean Francois Payen, MD, Principal Investigator — University Hospital, Grenoble
Locations (21):
- France (21):
  - CHRA Annecy, Annecy, Auvergne-Rhône-Alpes
  - CHU Grenoble, Grenoble, Isere
  - Ch Belley, Belley
  - CHU, Besançon
  - Ch Briancon, Briançon
  - Ch Cannes, Cannes
  - Ch Chambery, Chambéry
  - CHU, Clermont-Ferrand
  - CHU, Dijon
  - Ch Grasse, Grasse
  - Chu Edouard Herriot, Lyon
  - CHU Lyon, Lyon
  - CHU Pierre Benite, Lyon
  - CH Nantes, Nantes
  - Chu Nimes, Nîmes
  - Ch Saint Jean de Maurienne, Saint-Jean-de-Maurienne
  - Ch Saint Julien En Genevois, Saint-Julien-en-Genevois
  - Hopitaux Du Pays Du Mont Blanc, Sallanches
  - Ch Thonon Les Bains, Thonon-les-Bains
  - CH Valence, Valence
  - Ch Voiron, Voiron

REFERENCES:
- [Background] Thornhill S, Teasdale GM, Murray GD, McEwen J, Roy CW, Penny KI. Disability in young people and adults one year after head injury: prospective cohort study. BMJ. 2000 Jun 17;320(7250):1631-5. doi: 10.1136/bmj.320.7250.1631. PMID 10856063
- [Background] Davis DP, Kene M, Vilke GM, Sise MJ, Kennedy F, Eastman AB, Velky T, Hoyt DB. Head-injured patients who "talk and die": the San Diego perspective. J Trauma. 2007 Feb;62(2):277-81. doi: 10.1097/TA.0b013e31802ef4a3. PMID 17297312
- [Background] Livingston DH, Lavery RF, Passannante MR, Skurnick JH, Baker S, Fabian TC, Fry DE, Malangoni MA. Emergency department discharge of patients with a negative cranial computed tomography scan after minimal head injury. Ann Surg. 2000 Jul;232(1):126-32. doi: 10.1097/00000658-200007000-00018. PMID 10862205
- [Background] Marshall LF, Marshall SB, Klauber MR, van Berkum Clark M, Eisenberg HM, Jane JA, et al. A new classification of head injury based on computerized tomography. J Neurosurg 1991; 75: S14-S20.
- [Background] Wardlaw JM, Easton VJ, Statham P. Which CT features help predict outcome after head injury? J Neurol Neurosurg Psychiatry. 2002 Feb;72(2):188-92; discussion 151. doi: 10.1136/jnnp.72.2.188. PMID 11796768
- [Background] Sifri ZC, Homnick AT, Vaynman A, Lavery R, Liao W, Mohr A, Hauser CJ, Manniker A, Livingston D. A prospective evaluation of the value of repeat cranial computed tomography in patients with minimal head injury and an intracranial bleed. J Trauma. 2006 Oct;61(4):862-7. doi: 10.1097/01.ta.0000224225.54982.90. PMID 17033552
- [Background] af Geijerstam JL, Oredsson S, Britton M; OCTOPUS Study Investigators. Medical outcome after immediate computed tomography or admission for observation in patients with mild head injury: randomised controlled trial. BMJ. 2006 Sep 2;333(7566):465. doi: 10.1136/bmj.38918.669317.4F. Epub 2006 Aug 8. PMID 16895944
- [Background] Stein SC, Burnett MG, Glick HA. Indications for CT scanning in mild traumatic brain injury: A cost-effectiveness study. J Trauma. 2006 Sep;61(3):558-66. doi: 10.1097/01.ta.0000233766.60315.5e. PMID 16966987
- [Background] White H, Venkatesh B. Applications of transcranial Doppler in the ICU: a review. Intensive Care Med. 2006 Jul;32(7):981-94. doi: 10.1007/s00134-006-0173-y. Epub 2006 May 10. PMID 16791661
- [Background] McQuire JC, Sutcliffe JC, Coats TJ. Early changes in middle cerebral artery blood flow velocity after head injury. J Neurosurg. 1998 Oct;89(4):526-32. doi: 10.3171/jns.1998.89.4.0526. PMID 9761044
- [Background] Jaffres P, Brun J, Declety P, Bosson JL, Fauvage B, Schleiermacher A, Kaddour A, Anglade D, Jacquot C, Payen JF. Transcranial Doppler to detect on admission patients at risk for neurological deterioration following mild and moderate brain trauma. Intensive Care Med. 2005 Jun;31(6):785-90. doi: 10.1007/s00134-005-2630-4. Epub 2005 Apr 16. PMID 15834704
- See also: Username : DTC99 Password : DTCTST — https://www.clininfohosting.com/specif/DTC/